CLINICAL TRIAL: NCT02209519
Title: Randomized Controlled Trial of Treatment of Male Partners of Women With BV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, Jane Schwebke, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Bacterial Vaginosis
Keywords: bacterial vaginosis; recurrence; male partner
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole (Experimental): Male Partner: metronidazole 500 mg PO BID x 7days Female Partner: metronidazole 500 mg PO BID x 7days
  Interventions: Drug: Metronidazole (male partner)
- Placebo (Placebo Comparator): Male Partner: one tablet PO BID for 7 days Female Partner: metronidazole 500 mg PO BID x 7days
  Interventions: Other: Placeob (male partner)

INTERVENTIONS:
Drug: Metronidazole (male partner) — 500 mg PO BID for 7 days
  Arms: Metronidazole
Other: Placeob (male partner) — matching placebo capsules PO BID for 7 days
  Arms: Placebo

SUMMARY:
Male partners of womoen with recurrent bacteria vaginosis are randomized to treatment with metronidazole or placebo to compare the rates of recurrent BV in the women

DETAILED DESCRIPTION:
This study will be performed as a phase III randomized, double-blinded trial to evaluate the efficacy of 1) metronidazole 500 mg PO BID for 7 days versus 2) placebo capsules alone for treatment of the male sexual partner of women with recurrent BV. The primary outcome is the rates of recurrent BV between these two groups. Although this is a phase III study we will carefully monitor potential toxicity in the males since it is currently not standard of care to treat males for this indication.

Women with symptomatic BV defined by Amsel criteria 1 and no evidence of STD will be invited to participate. Inclusion criteria are that the woman be at least 18 years of age, heterosexual, have symptoms of vaginal odor and/or discharge, meet the modified clinical (Amsel) criteria for BV (all must have a vaginal pH of >4.5, a positive whiff test, and clue cells to be eligible), have an enrollment Nugent score of 7 or greater, and a history of 2 or more episodes of BV in the previous year. She must have a regular current sex partner who would be willing to participate. We will exclude women who have had recurrent BV for greater than 3 years as well as women who have failed previous treatment studies since it is likely that these women are having recurrent BV as a result of relapse of the BV biofilm as opposed to reinfection.

Follow-up visits will be conducted at day 21, 8 and 16 weeks. At each follow-up visit, a questionnaire will be administered, diary reviewed, pelvic examination conducted and specimens (Gram stain, Amsel criteria, G vaginalis culture and detection of novel organisms) obtained as done at the enrollment visit. Participants will be asked to return the medication packages, a standard way of assessing adherence to the regimen. Cure will be ascertained using the clinical criteria for BV of Amsel 1 as well as the Nugent scoring system 16. The persistence or disappearance of specific organisms will be analyzed in relationship to these standard definitions of cure. Women who fail initial therapy or have recurrence of symptomatic BV during the course of the study will be re-treated with 7 days of metronidazole and dropped from the study at that time. Any woman found to have a positive screening test for gonorrhea or chlamydia will be treated appropriately and instructed to notify her partner of the need to be treated. Women with intercurrent vaginal yeast infections, which may occur, will be treated with oral fluconazole and continued in the study. Women with a positive culture for trichomonas will be dropped from the study as their male partners will require treatment with metronidazole.

Male Study Procedures

Males referred by their female sexual partner will be seen within 48 hours of enrollment of the female. Males will be consented and asked behavioral and historical questions using a gender appropriate questionnaire, with special emphasis on number of current sexual partners. A couple verification screening tool will be utilized to be certain they are current sexual partners48. The confidentiality of their answers will be emphasized. They will be examined and a urethral swab specimen obtained to be used for G vaginalis culture and then archived. Following the swabs, two external swabs from the coronal sulcus and a 10 ml first void urine specimen will be obtained. These specimens will also be used for G vaginalis culture and archived for possible use in detection of novel organisms. The urine will also be used for NAATS for N gonorrhoeae and C trachomatis and for the determining the presence or absence of Gardnerella biofilm24. They will then be randomized to one of two treatment arms:

1. Metronidazole 500 mg PO twice a day for 7 days .
2. Placebo capsules PO twice a day for 7 days.

Both arms will also contain an instruction sheet on metronidazole.

ELIGIBILITY:
Inclusion Criteria: Female

1. At least 18 years of age (19 years of age in Alabama due to State law)
2. Sexual partner to a female who meets study eligibility
3. Willingness to provide informed consent
4. Willingness to abstain from sexual intercourse or use condoms {during the study}
5. Willingness to abstain from alcohol for the first week of the study

Inclusion Criteria: Male

1. At least 18 years of age (19 years of age in Alabama due to State law)
2. Heterosexual with a regular partner
3. History of 2 or more episodes of BV in the previous 12 months
4. Symptoms of BV including vaginal discharge and/or odor
5. Positive Amsel criteria for BV including vaginal pH >4.5, positive whiff test, presence of clue cells
6. Willingness to provide informed consent
7. Willingness to abstain from sexual intercourse or use condoms {during the study}
8. Willingness to abstain from alcohol for the first week of the study

Exclusion criteria (both genders)

1. Allergy to metronidazole
2. Failure of the male partner to keep his appointment to be seen within 48 hours
3. Pregnant or breast feeding (females)
4. HIV or other chronic disease which in the opinion of the investigator would interfere with the ability to participate in this study
5. Subject requires concurrent lithium, coumadin, dilantin, or antabuse
6. Presence of trichomonas on wet prep of vaginal fluid (females)
7. Women with a history of recurrent BV for >3 years or women who have failed previous treatment studies for BV

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jane Schwebke, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jane Schwebke, Pell City, Alabama, United States

REFERENCES:
- [Derived] Schwebke JR, Lensing SY, Lee J, Muzny CA, Pontius A, Woznicki N, Aguin T, Sobel JD. Treatment of Male Sexual Partners of Women With Bacterial Vaginosis: A Randomized, Double-Blind, Placebo-Controlled Trial. Clin Infect Dis. 2021 Aug 2;73(3):e672-e679. doi: 10.1093/cid/ciaa1903. PMID 33383580

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Male Partner: one tablet PO BID for 7 days Female Partner: metronidazole 500 mg PO BID x 7days
  Placebo (male partner): matching placebo capsules PO BID for 7 days
Period: Overall Study
Arm/Group | Metronidazole | Placebo
Started | 107 | 107
Completed | 107 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Placebo | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (6.9) | 32.8 (8.1) | 32.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 14 | 15 | 29
  african american | 89 | 88 | 177
  multiracial | 4 | 4 | 8
  hispanic | 6 | 4 | 10
  non-hispanic | 101 | 103 | 204
Region of Enrollment [Number; unit: participants]
  United States | 107 | 107 | 214

OUTCOME MEASURES:

1. Primary Outcome: Number of Female Partners Whose Male Partners Received Metronidazole Versus Females Whose Male Partners Did Not Receive Metrodiazole With Recurrence of BV in the Female
Description: the female partners will be assessed for recurrence/persistence of BV. tRecurrence/persistence is measured by - Positive 3 - 4 Amsel criteria (vaginal pH > 4.7, clue cells, positive whiff test, homogenous discharge); Nugent score >3
  No Recurrence/Persistence is measured by:
  - Presence of 0 -2 Amsel criteria; Nugent score 0-3.
Time Frame: 16 weeks post start of receipt of study drug
Population: those completing the study
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 107 | 107
Participants | 87 | 86

2. Secondary Outcome: Time to Recurrence of BV in Women Whose Partner Received Metronidazole Versus Females Whose Partners Did Not Receive Metronidazole
Description: time to recurrence measured in days
Time Frame: from the end of week 1 up to 16 weeks
Population: unable to collect data due to lab issues
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline through 16 weeks
Arm/Group | Metronidazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107 | 1/107
Other Adverse Events (participants affected / at risk) | 29/107 | 31/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metronidazole (N=107) | Placebo (N=107)
trauma (Musculoskeletal and connective tissue disorders) | 0 | 1 — motor vehicle accident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=107) | Placebo (N=107)
Infections and infestations (Infections and infestations) | 18 (18) | 21 (21)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
musculoskelatal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
nervous (Nervous system disorders) | 1 (1) | 3 (3)
psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
reproductive system (Reproductive system and breast disorders) | 1 (1) | 0 (0)
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
gastrointestinal (Gastrointestinal disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT02209519/Prot_SAP_000.pdf